CLINICAL TRIAL: NCT05618210
Title: Comparison of the Effect of ESPB and Rhomboid Block on Postoperative Pain and Opioid Consumption in Patients Undergoing Lobectomy With VATS Method: a Randomized Controlled Study
Brief Title: Effect of ESPB and Rhomboid Block on VATS Method
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, assistant professor, Marmara University
Other Study IDs: 09.2022.756
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Opioid Consumption; Postoperative Pain; Complication,Postoperative
Keywords: ESPB; RHOMBOİD BLOCK; OPİOİD; POSTOPERATİVE PAIN
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- erector spinae plane block group: In the ESPB group, after the patients are placed in the prone position, the linear ultrasound probe will be placed in the midline in the transverse plane to visualize the spinous processes, and the transverse process, trapezius, latissimus dorsi and erector spina muscles will be visualized on the side where VATS is planned at the T5 vertebra level. With an 'in-plane' approach, using a 22 gauge 5-8 cm block needle with extension line (Braun, Melsungen, Germany), which can be seen on ultrasound, the skin, subcutaneous and trapezius, latissimus dorsi and erector spina muscles are passed in the cranio-caudal direction and 0.5- After confirming the needle site with 1 ml of saline, the ESPB will be administered with 20 ml of 0.5% bupivacaine by visualizing the local anesthetic spread linearly.
  Interventions: Other: regional anesthesia
- Rhomboid block: In the rhomboid intercostal block group, after the patients are placed in the prone position, the ipsilateral arm is positioned towards the chest, allowing the scapula to move laterally and the area called auscultation triangle to be opened, and after the skin disinfection of the surgical side; By using a linear ultrasound probe, the rhomboid major and intercostal muscles will be defined in the auscultation triangle region, and a 50-80 mm needle will be injected into the plan between them at the T5-6 level with an in-plane approach with 20 ml of 0.5% bupivacaine and local anesthetic injection.
  Interventions: Other: regional anesthesia

INTERVENTIONS:
Other: regional anesthesia — in the ESPB group, the linear ultrasound probe was placed in the erector spina muscles were visualized on the side where VATS was planned. block needle can be seen on ultrasound, the skin and erector spina muscles are passed in the cranio-caudal direction. ESPB will be administered with 20 ml of 0.5% bupivacaine by visualizing the local anesthetic spread linearly.
  In the rhomboid intercostal block group, the ipsilateral arm is positioned towards the chest, allowing the scapula to move laterally and the area called auscultation triangle to be opened, and after the skin disinfection of the surgical side; By using a linear ultrasound probe, the rhomboid major and intercostal muscles will be defined in the auscultation triangle region, and T5-6 level with an in-plane approach with 20 ml of 0.5% bupivacaine and local anesthetic injection.

SUMMARY:
The aim of this study is to compare ultrasound-guided ESBP and Rhomboid block in terms of postoperative pain management, postoperative opioid consumption and complications in patients undergoing lobectomy with VATS.Patients aged 18-75 years, ASA 1-2-3, who gave informed consent to lobectomy with video-assisted thoracic surgery (VATS) method will be included in this study. Patients with contraindications for the application of either method, known chronic pain, local anesthetic allergy, spinal deformity or mental or psychiatric problems that prevent cooperation, taking anticoagulants, and infection at the injection site will not be included in the study. Patients who agree to participate in the study will be randomly assigned to one of the anesthesia groups of the study, which include ESPB (elector spina plane block) (Group 1) or Rhomboid block (Group 2). Randomization will be at a ratio of 1:1 and will be done by the closed-envelope method. Beforehand, a piece of paper with the name of one of the two groups will be placed inside the envelopes and the envelopes will be closed and mixed. A closed envelope will be drawn randomly for each patient before the procedure, and procedures will be carried out according to the group specified on the paper.

DETAILED DESCRIPTION:
Video-assisted thoracic surgery (VATS); Although it causes less postoperative pain compared to traditional thoracotomy, it can still cause significant postoperative problems. Relief of postoperative pain; it eliminates the undesirable pathological effects of pain, reduces the length of hospital stay and costs. Thoracic epidural analgesia and paravertebral block are recommended for the relief of postoperative pain after thoracotomy. Bendixen et al. Because VATS is less painful; recommended less invasive regional techniques and systemic analgesics. For the relief of postoperative pain after VATS; paravertebral block, erector spina plan block (ESPB), and serratus plan block have been successfully applied. In order to provide analgesia after VATS; the most appropriate techniques or protocols need to be determined. ESPB; In 2016, Forero et al. and is used for the control of pain after many surgical procedures. ESPB has been successfully applied for the relief of postoperative pain after VATS. Elsharkawy et al. have shown that rhomboid intercostal block can be beneficial in providing adequate analgesia for both anterior and posterior hemithorax, in cadaver studies, but it is better with methods that are useful in relieving pain after VATS previously. They say more comparisons are needed. In recent studies, it has been shown that rhomboid intercostal block is effective in relieving postoperative pain in comparison with control groups. More randomized controlled studies are needed to demonstrate that rhomboid intercostal block provides effective analgesia in VATS. The aim of this study is to compare ultrasound-guided ESBP and Rhomboid block in terms of postoperative pain management, postoperative opioid consumption and complications in patients undergoing lobectomy with VATS.

The aim of this study is to compare ultrasound-guided ESBP and Rhomboid block in terms of postoperative pain management, postoperative opioid consumption and complications in patients undergoing lobectomy with VATS.Patients aged 18-75 years, ASA 1-2-3, who gave informed consent to lobectomy with video-assisted thoracic surgery (VATS) method will be included in this study. Patients with contraindications for the application of either method, known chronic pain, local anesthetic allergy, spinal deformity or mental or psychiatric problems that prevent cooperation, taking anticoagulants, and infection at the injection site will not be included in the study. Patients who agree to participate in the study will be randomly assigned to one of the anesthesia groups of the study, which include ESPB (elector spina plane block) (Group 1) or Rhomboid block (Group 2). Randomization will be at a ratio of 1:1 and will be done by the closed-envelope method. Beforehand, a piece of paper with the name of one of the two groups will be placed inside the envelopes and the envelopes will be closed and mixed. A closed envelope will be drawn randomly for each patient before the procedure, and procedures will be carried out according to the group specified on the paper.

Intraoperative anesthesia management The patients in this group were on the operating table before induction of anesthesia, and in the ESPB group (Group 1), after the patients were placed in the prone position, the linear ultrasound probe was placed in the midline in the transverse plane, and spinous processes were visualized at the T5 vertebra level, and the transverse process, trapezius, latissimus dorsi and erector spina muscles were visualized on the side where VATS was planned. will be displayed. With an 'in-plane' approach, using a 22 gauge 5-8 cm block needle with extension line (Braun, Melsungen, Germany), which can be seen on ultrasound, the skin, subcutaneous and trapezius, latissimus dorsi and erector spina muscles are passed in the cranio-caudal direction and 0.5- After confirming the needle site with 1 ml of saline, the ESPB will be administered with 20 ml of 0.5% bupivacaine by visualizing the local anesthetic spread linearly.

In the rhomboid intercostal block group (Group 2), after the patients are placed in the prone position, the ipsilateral arm is positioned towards the chest, allowing the scapula to move laterally and the area called auscultation triangle to be opened, and after the skin disinfection of the surgical side; By using a linear ultrasound probe, the rhomboid major and intercostal muscles will be defined in the auscultation triangle region, and a 50-80 mm needle will be injected into the plan between them at the T5-6 level with an in-plane approach with 20 ml of 0.5% bupivacaine and local anesthetic injection.

Under standard monitoring (ECG, non-invasive blood pressure, and finger oxygen saturation), anesthesia induction will be performed with propofol (2 mg/kg), remifentanil 1mcg/kg, and rocuronium 0.6 mg/kg. Bispectral index (BIS) and analgesia nociception index (ANI) monitoring will be started immediately after intubation. Anesthesia will be maintained with remifentanil infusion, with ANI > 50 and BIS < 50. Patients were given 1 g i.v. before waking up after surgery. paracetamol will be given. Measurements Perioperative clinical and demographic data of each patient will be collected: age, gender, diagnosis, operation, ASA, duration of surgery, duration of anesthesia. Intraoperatively, heart rate, blood pressure, ANI and BIS measurements will be made and recorded in all patients at 15-minute intervals. The total intraoperative opioid dose will also be recorded.

Post-awakening pain will be assessed and recorded using the visual analog scale (VAS), then patient-controlled analgesia (PCA) will be initiated, with all patients locked in 15 minutes and given 4 mg of morphine at each application by the patient. Pain assessment will be done with VAS at 6, 12, 24 and 48 hours postoperatively. In the postoperative period, the amount of morphine administered by PCA (in the first and second 24 hours) and any additional analgesics required (tramadol, paracetamol, etc.) will be recorded.

sample size In a previous study, based on the consumption of morphine equivalent in the first 24 hours (approximately 2.75 mg standard deviation) [8], it was found that 33 patients per group were required to detect the 2.5 mg difference between the two groups with 90% power and 5% alpha error. . Considering that there may be a dropout of approximately 10 percent, it is planned to include at least 35 patients in each group.

Statistical analysis In the comparison of the two groups in terms of continuous numerical variables, Student t test or Mann-Whitney U test will be used for independent samples according to distribution. Groups will be compared in terms of categorical variables using the Pearson chi-square test or the Fisher exact test. Two-way ANOVA test will be used for repeated measurements in comparison of groups in terms of the course of postoperative VAS scores and intraoperative heart rate, blood pressure, ANI, BIS variables over time. A value of p<0.05 will be accepted as an indicator of significance in the tests.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-75 years, ASA 1-2-3 who gave informed consent

Exclusion Criteria:

Patients with contraindications, known chronic pain, local anesthetic allergy, spinal deformity or mental or psychiatric problems that prevent cooperation, taking anticoagulants, infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 years, ASA 1-2-3 who gave informed consent
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
postoperative pain management | postoperatif first 24 hours.
  record of postoperative visual analog scala 0-10 values

SECONDARY OUTCOMES:
opioid consumption | postoperatif first 24 hours.
  record of postoperative opioid consumption with patients control device

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)